CLINICAL TRIAL: NCT03488212
Title: Pragmatic Trial of Technology-Supported Behavioral Obesity Treatment in the Primary Care Setting: A Multiphase Effectiveness and Implementation Hybrid Design
Brief Title: Online Obesity Treatment in Primary Care (Rhode Island, USA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John Graham Thomas, Associate Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18DK114715 (NIH); R18DK114715 (NIH)
Record Dates: First submitted 2018-03-22; First posted 2018-04-04 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Basic Implementation Intervention (Active Comparator)
  Interventions: Behavioral: Training to Identify Eligible Patients and Direct them to Online Obesity Treatment Program
- Enhanced Implementation Intervention (Experimental)
  Interventions: Behavioral: Training to Identify Eligible Patients and Direct them to Online Obesity Treatment Program; Behavioral: Training to Motivate and Support Patients' Weight Loss
- Online Treatment; Control Maintenance Intervention (Active Comparator)
  Interventions: Behavioral: Online Behavioral Weight Loss Intervention; Behavioral: Control Intervention for Weight Loss Maintenance and Weight Gain Prevention
- Online Treatment; Monthly Lessons & Feedback for Maintenance (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Intervention; Behavioral: Monthly Lessons and Feedback Intervention for Weight Loss Maintenance and Weight Gain Prevention
- Online Treatment; Refresher Courses for Maintenance (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Intervention; Behavioral: Refresher Courses for Weight Loss Maintenance and Weight Gain Prevention

INTERVENTIONS:
Behavioral: Training to Identify Eligible Patients and Direct them to Online Obesity Treatment Program — Primary care clinic staff are trained to identify patients who meet study inclusion and exclusion criteria. They are then trained to provide patients with the information necessary to enroll in the study and access the online behavioral obesity treatment.
  Arms: Basic Implementation Intervention; Enhanced Implementation Intervention
Behavioral: Training to Motivate and Support Patients' Weight Loss — Primary care clinic staff are trained in psychological and behavioral strategies for: talking to patients about weight and weight loss in a way that patients find acceptable and helpful, increasing motivation for weight loss, overcoming common barriers to weight loss, and persevering with a weight loss attempt. They are trained in strategies to provide this support by telephone in addition to during clinic visits.
  Arms: Enhanced Implementation Intervention
Behavioral: Online Behavioral Weight Loss Intervention — For 3 months, participants receive: a weekly online lessons for training in behavioral skills for losing weight; online self-monitoring of daily weight, diet, and physical activity; weekly feedback on the self-monitoring record.
  Arms: Online Treatment; Control Maintenance Intervention; Online Treatment; Monthly Lessons & Feedback for Maintenance; Online Treatment; Refresher Courses for Maintenance
Behavioral: Control Intervention for Weight Loss Maintenance and Weight Gain Prevention — After completing the 3-month Online Behavioral Weight Loss Intervention, participants receive 9 months of: monthly online newsletters with educational information pertaining to healthy weight, diet, and physical activity habits.
  Arms: Online Treatment; Control Maintenance Intervention
Behavioral: Monthly Lessons and Feedback Intervention for Weight Loss Maintenance and Weight Gain Prevention — After completing the 3-month Online Behavioral Weight Loss Intervention, participants receive 9 months of: monthly online lessons for training in behavioral skills for maintaining weight loss and preventing weight gain; online self-monitoring of daily weight, diet, and physical activity; monthly feedback on the self-monitoring record.
  Arms: Online Treatment; Monthly Lessons & Feedback for Maintenance
Behavioral: Refresher Courses for Weight Loss Maintenance and Weight Gain Prevention — After completing the 3-month Online Behavioral Weight Loss Intervention, participants receive two month-long refresher courses with weekly online lessons for training in behavioral skills for maintaining weight loss and preventing weight gain; online self-monitoring of daily weight, diet, and physical activity; weekly feedback on the self-monitoring record; weekly challenges focuses on specific behavior change and weight loss goals.
  Arms: Online Treatment; Refresher Courses for Maintenance

SUMMARY:
Behavioral obesity treatment produces clinically significant weight loss; for the greatest impact, it should be made available in the primary care setting where it can reach the many patients with overweight/obesity. The investigators developed a 3-month automated online behavioral weight loss program, Rx Weight Loss (RxWL), and showed that it produces clinically significant weight losses among primary care patients. The investigators' early efforts at pragmatic implementation of RxWL have been promising, and have shed light on challenges associated with implementation, and the need to study longer-term effectiveness. The investigators will therefore conduct a pragmatic study to improve the implementation and effectiveness of this behavioral obesity intervention delivered in routine and representative healthcare settings. The investigators are partnering with the Rhode Island Primary Care Physicians Corporation (RIPCPC), a large primary care network of 58 practices with 100 physicians and 16 nurse care managers. Using the framework for Effectiveness-Implementation Hybrid Designs, the investigators will simultaneously target effectiveness and implementation to maximize the public health impact of the research. Half of the 16 nurse care managers, and the practices they serve, will be randomized to either Basic Implementation (alerts generated using the electronic medical record [EMR] to direct eligible patients to RxWL), or to the Enhanced Implementation (alerts, clinician skills training to motivate and support weight loss, clinician dashboard with reports on patient progress and tools to facilitate patient engagement and behavior change). The investigators will test the hypothesis that the Enhanced Implementation will increase the proportion of patients directed to, enrolling, and completing the weight loss program. Because maintenance of weight loss is a critical problem, this project will also involve randomization of 600 patients with overweight/obesity and type 2 diabetes, hypertension, and/or hypercholesterolemia to the 3 month RxWL intervention followed by one of three maintenance conditions: (a) Control- 9 monthly online education sessions; (b) Monthly Lessons and Feedback- 9 monthly online video lessons teaching self-regulation with automated feedback on the self-monitoring record; (c) Refresher Campaigns- 9 monthly on-line video sessions, teaching self-regulation and providing two 4-week courses with novel strategies and behavioral challenges to improve long-term outcomes. The investigators will test the hypothesis that 12-month weight losses are better with Refresher Campaigns than Monthly Lessons and Feedback, and both are better than Control. Secondary outcomes include changes in weight, CVD risk factors, and medication use over a full 24 months. The project is significant and innovative because: it uses an empirically validated approach to obesity treatment that is integrated into the primary care setting, leveraging existing staff and EMR capabilities; it has a dual focus on improving effectiveness and implementation; it has a pragmatic design in partnership with a large primary care network that treats a diverse patient population; and it has potential to it provides a scalable, sustainable approach that can serve as a model for broader dissemination of obesity treatment intervention.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25-45 kg/meters-squared
* one or more cardiovascular risk factor (type 2 diabetes, hypercholesterolemia, or hypertension)

Exclusion Criteria:

* currently in another active weight loss program
* taking weight loss medication
* currently pregnant, lactating
* <6 months post-partum
* plan to become pregnant during the next 12 months
* a medical condition that would affect the safety of participating in unsupervised physical activity
* inability to walk 2 blocks without stopping

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Weight | 12 months after study enrollment

SECONDARY OUTCOMES:
Change in Weight | 24 months after study enrollment
Proportion of Patients Achieving a Weight Loss of ≥5% of Initial Body Weight | 12 and 24 months after study enrollment
Patient Satisfaction with the Treatment Program | 3 and 12 months after study enrollment
  Using a questionnaire developed for this study, patients are asked to rate their overall satisfaction with the treatment program, specific components of the treatment program, and the likelihood that they would recommend the program to family and friends, on a 5-point Likert scale ranging from 1 (Low) to 5 (High).
Provider Satisfaction with the Treatment Program | 12 months after study enrollment
  Using a questionnaire developed for this study, providers are asked to rate their overall satisfaction with the treatment program, and specific components of the treatment program, on a 5-point Likert scale ranging from 1 (Low) to 5 (High).
Proportion of Patients Deemed Eligible by the Electronic Medical Record Who are Directed to the Online Treatment Program | 24 months after study initiation
  The proportion of patients who approached by clinic staff for potential participation in the study, out of the patients who are deemed potentially eligible in reports generated using the electronic medical record.
Proportion of Patients That Enroll After Being Directed to the Online Treatment Program | 24 months after study initiation
  The proportion of patients who enroll in the study out of the patients who are approached by clinic staff for potential participation in the study.
Proportion of Enrolled Patients who Complete the Online Treatment Program | 24 months after study initiation
  The proportion of patients who complete the initial 3-month weight loss treatment and following 9-month weight loss maintenance and weight gain prevention program, out of those that enroll.
Clinician Contact with Patients Directed to the Online Treatment Program | 24 months after study initiation
  Number and type of clinician contact with patients (e.g., clinic visits, phone calls).
Patient Engagement and Adherence to the Online Intervention. | 12 months after study enrollment
  The online treatment platform automatically records all aspects of use including logins, lessons viewed, and self-monitoring records submitted.
Clinician Engagement with the Online Treatment Platform | 24 months after study initiation
  Frequency and type of use (e.g., viewing patients progress metrics) of the online platform for tracking patient progress in the online treatment.
Change in Low-density Lipoprotein (mg/dL) | 12 and 24 months after study enrollment
Change in High-density Lipoprotein (mg/dL) | 12 and 24 months after study enrollment
Change in Triglycerides (mg/dL) | 12 and 24 months after study enrollment
Change in Blood Glucose (mg/dL) | 12 and 24 months after study enrollment
Change in Glycated Haemoglobin (HbA1c) | 12 and 24 months after study enrollment
Change in Systolic Blood Pressure (mmHG) | 12 and 24 months after study enrollment
Change in Diastolic Blood Pressure (mmHG) | 12 and 24 months after study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Graham Thomas, PhD, Principal Investigator — The Miriam Hospital; Rena R Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control and Diabetes Resarch Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas JG, Panza E, Goldstein CM, Hayes JF, Benedict N, O'Leary K, Wing RR. Pragmatic Implementation of Online Obesity Treatment and Maintenance Interventions in Primary Care: A Randomized Clinical Trial. JAMA Intern Med. 2024 May 1;184(5):502-509. doi: 10.1001/jamainternmed.2023.8438. PMID 38466266
- [Derived] Thomas JG, Panza E, Espel-Huynh HM, Goldstein CM, O'Leary K, Benedict N, Puerini AJ, Wing RR. Pragmatic implementation of a fully automated online obesity treatment in primary care. Obesity (Silver Spring). 2022 Aug;30(8):1621-1628. doi: 10.1002/oby.23502. PMID 35894075